CLINICAL TRIAL: NCT01891214
Title: Validation of the French Version of the Inflammatory Bowel Disease Questionnaire (IBDQ) for Ulcerative Colitis and Crohn's Disease
Acronym: F-IBDQ
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00144-41; LOC/12-17 Bouguen F-IBDQ (Other: Rennes University Hospital)
Record Dates: First submitted 2013-06-17; First posted 2013-07-03 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Inflammatory bowel diseases; Inflammatory Bowel Disease Questionnaire (IBDQ)
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ulcerative Colitis and Crohn's Disease
  Interventions: Other: Validation of the French Version of the Inflammatory Bowel Disease Questionnaire (IBDQ)

INTERVENTIONS:
Other: Validation of the French Version of the Inflammatory Bowel Disease Questionnaire (IBDQ)

SUMMARY:
The purpose of the study is to develop a validated French version of the IBDQ in a cohort of patients suffering from Inflammatory bowel diseases, namely Crohn's disease and Ulcerative Colitis.

DETAILED DESCRIPTION:
Importance of measuring subjective aspects of the patient's health, often referred to as quality of life (QoL), become increasingly recognized and integrated into healthcare. For this purpose, The Inflammatory Bowel Disease Questionnaire (IBDQ) is a widely used questionnaire for QoL assessment specific for patients who suffer from inflammatory bowel diseases. However, the IBDQ was originally developed in a cohort of Canadian patients in English language. Since QoL is impacted by underlying cultural trends, any translation of the IBDQ should be reassessed in relation to its validity, reliability, and sensitivity to detect change in the new language and cultural context. While the linguistic French translation of the original IBDQ has been validated, the French IBDQ has never been tested adequately on a French cohort of patient that we aim to perform.

ELIGIBILITY:
Inclusion Criteria:

* men and women ≥ 18 years of age,
* patient with definite diagnosis of UC or CD for at least 6 months

Exclusion Criteria:

* adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty
* inability to comprehend or complete the self-administered questionnaire
* psychiatric diagnosis that prevents participation (many pts will have anxiety or depression and should not be excluded)
* stoma
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with definite diagnosis of UC or CD for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Internal validity, scale F-IBDQ | Day1 and Month4
  Chronbach's alpha coefficient, measured at the first visit and at the second visit.
External validity, questionnaire SF36 | Day1 and Month4
  Correlation with the French validated SF-36 and disease activity indexes (Harvey Bradshaw index for Crohn's disease and Simple Colitis Activity Index for ulcerative colitis, measured at the first visit and at the second visit.
Discriminant ability, disease activity indexes | Day1 and Month4
  Correlation with disease activity indexes, measured at the first visit and at the second visit.
Reliability, disease outcomes | Day1 and Month4
  Correlation with disease outcomes, measured at the first visit and at the second visit.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Bouguen, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - CHRU de Nancy, Nancy
  - Service des Maladies de l'Appareil Digestif, Hôpital de Pontchaillou, 2 rue Henri Le Guilloux, Rennes